CLINICAL TRIAL: NCT01499459
Title: Efficacy of Exvivo Expanded Autologous Mesenchymal Stem Cell Transplantation Via Peripheral Vein in Patients With Liver Cirrhosis
Brief Title: Autologous Mesenchymal Stem Cell Transplantation in Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Murat Kantarcioglu, Gulhane Military Medical Academy, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11111111; 1111111 (Other: Gulhane School of Medicine)
Record Dates: First submitted 2011-12-14; First posted 2011-12-26 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; autologous mesenchymal stem cell transplantation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous mesenchymal stem cell transplantation (Experimental)
  Interventions: Genetic: autologous mesenchymal stem cell transplantation

INTERVENTIONS:
Genetic: autologous mesenchymal stem cell transplantation — Every patient is given 1x106 MSCs per kg infused via peripheral vein.

SUMMARY:
This study is aiming to investigate the efficacy of autologous mesenchymal stem cell (MSC) transplantation in 25 randomized patients with liver cirrhosis autologous mesenchymal stem cell will be derived from patients' bone marrows and will be infused via peripheral vein. Liver biopsies will be performed in every patient in the beginning and at 6th month.

ELIGIBILITY:
Inclusion Criteria:

* radiological, clinical and histopathological diagnosis of liver cirrhosis
* absence of hepatocellular carcinoma or any malignancies
* no psychiatric disorder
* no serous cardiovascular and pulmonary comorbidities
* serum total bilirubin levels less than 5 mg/dL
* platelet counts more than 30.000 mm3
* more than one year follow up period after initiation of antiviral drugs

Exclusion Criteria:

* alcohol intake in last one year
* initiation of antiviral medication in last one year
* systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
clinical improvement | clinical improvement parameters will be assessed six month after mesenchymal stem cell transplantation
  biochemical and hematologic parameters

SECONDARY OUTCOMES:
liver regeneration | 6.th month after MSC transplantation
  histopathologic assesments comparing before and at 6th month liver biopsies

CONTACTS AND LOCATIONS:
Overall Officials: murat kantarcioglu, MD, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- Gulhane Military Medical Academy Department of Gastroenterology, Ankara, Turkey (Türkiye)